CLINICAL TRIAL: NCT00683566
Title: State Dependent Resonance in the BG-cortical Loops
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2007-A01178-45; 2007 36
Record Dates: First submitted 2008-02-26; First posted 2008-05-23 (Estimated); Last update posted 2014-08-28 (Estimated); Status verified 2014-08

CONDITIONS: Parkinson Disease
Keywords: parkinson
MeSH Terms: conditions — Parkinson Disease | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): A session in condition ON DOPAMINE and the other one in condition OFF DOPAMINE.
  Interventions: Procedure: electrostimulation

INTERVENTIONS:
Procedure: electrostimulation — Stimulate STN (at 0, 5, 10, 15, 20, 25, 30, 40, 70 and 130 Hz) in chronically implanted patients at rest and during simple and complex motor tasks

SUMMARY:
Neuronal activity in circuits between the basal ganglia (BG) and motor cortical areas is abnormally synchronized and rhythmic. The oscillatory activity prevails at 8-30 Hz in untreated Parkinson's Disease (PD) and its amplitude at both subthalamic and cortical levels inversely correlates with motor impairment. Moreover, these different levels in BG-cortical loops are coherent in this frequency band. The 8-30 Hz activity is suppressed by treatment following treatment with dopaminergic drugs and is partially suppressed prior to and during voluntary movements. An unanswered question is how do BG-cortical loops become so prominently engaged in this oscillatory activity? One possible explanation is that the resonance frequencies of the loops fall in the 8-30 Hz band in the untreated state, so that oscillations in this band are transmitted particularly well. So we hypothesize loop resonances in the 8-30 Hz frequency band at rest, which should be suppressed during movement and following dopaminergic therapy.

DETAILED DESCRIPTION:
Stimulate STN (at 0, 5, 10, 15, 20, 25, 30, 40, 70 and 130 Hz) in chronically implanted patients at rest and during simple and complex motor tasks while recording the steady state evoked potential over the cortex using EEG over the 19 sites of the classical 10/20 system and a channel to record artifact over the stimulator. Experiments will be carried out both in the OFF medication and ON medication condition.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease idiopathic evolving for more than 5 years
* Electrodes of stimulation implanted in 2 nuclei under - thalamic in the service of functional and stereotaxic neurosurgery of the CHU La timone for at least 6 months
* Doped sensibility superior to 50 % (estimated by the section III of the score UPDRS)
* Efficiency of the stimulation superior to 30 % (estimated by the section III of the score UPDRS)

Exclusion Criteria:

* Patients not verifying the criteria of inclusion
* Absence of data concerning the location of electrodes

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-02; Primary Completion 2010-02 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
The results are expected to bring further light into the understanding of the mechanisms underlying the propagation of pathological oscillatory activities in PD and may provide a basis for different therapeutic strategies. | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: jean philippe AZULAY, MD, Principal Investigator — AP-HM
Locations (1):
- AP-HM Timone, Marseille, Bouches Du Rhone, France